CLINICAL TRIAL: NCT06168227
Title: A Multicenter and Real-world Analysis of Clinical Outcomes and Safety of the Novel Recombinant Humanized Anti-HER2 Therapeutic Antibody RC48-ADC in Patients With HER2-positive or HER2-low Expressing, Locally Advanced or Metastatic Breast Cancer
Brief Title: A Multicenter and Real-world Analysis of RC48-ADC in Patients With HER2-positive or HER2-low Expressing, Locally Advanced or Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 20230905RC48
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Breast Cancer
Keywords: HER2-positive; HER2-low; ADC; RC48
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Patients receive RC48
  Interventions: Drug: Disitamb Vedotin

INTERVENTIONS:
Drug: Disitamb Vedotin — RC48-ADC based therapy
  Other Names: RC48

SUMMARY:
Evaluate the efficacy and safety of Disitamb Vedotin in patients with HER2-positive or HER2-low expressing, locally advanced or metastatic breast cancer

DETAILED DESCRIPTION:
The main goal of this clinical trial is to examinie the utilization of RC48 in different HER2 statuses, elucidating its clinical outcomes and safety, and investigating the factors that influence its clinical efficacy. The primary endpoint was the objective response rate (ORR) assessed by the primary researcher. Secondary endpoints included progression-free survival (PFS), overall survival (OS), disease control rate (DCR), time to progression, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. histopathologically or imaging-confirmedlocally advanced or metastatic breast cancer ;
2. HER2-positive or low status;
3. the function of major organswas normal, no treatmentcontraindications , andthe estimated survival time was more than 2 months;
4. at least one extracranialmeasurable lesion or osteolytic or mixed bone metastases inaccordance with the Response Evaluation Criteria in Solid Tumors v. 1.1 (RECIST 1.1);
5. the clinical data were complete and traceable.

Exclusion Criteria:

1. age <18 ye ars old;
2. other concurrent cancers;
3. patients who rece ived RC48 as a neoadjuvant or adjuvant regimen；
4. Incomplete medical data.

Ages: 18 Years to 85 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with HER2-positive or HER2-low expressing, locally advanced or metastatic breast cancer were eligible and received RC48 2.5 mg/kg every two weeks alone or combined with drugs with different anti-tumor mechanisms, such as immune checkpoint inhibitors (ICIs), tyrosine kinase inhibitors (TKIs) and antiangiogenic compounds.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
Objective Response Rate (ORR) | 2 years
  The overall response rate is defined as the percentage of patients with a best overall response of CR or PR relative to the appropriate analysis set

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Adverse Events (AE) | 2 years
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).
Overall Survival (OS) | 2 years
  It is defined as the time from the start of treatment to death for any reason.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No